CLINICAL TRIAL: NCT00491504
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study Using Subjective and Objective Measures to Evaluate the Clinical Efficacy of Mometasone Furoate Nasal Spray (MFNS) Following Initial and Maintenance Dosing in Subjects With Allergen-Induced Seasonal Allergic Rhinitis (SAR) in an Environmental Exposure Chamber (EEC)
Brief Title: This Study Contains an Active Drug Treatment Group With Mometasone Furoate Nasal Spray and a Placebo (Dummy) Treatment Group for Seasonal Allergic Rhinitis (SAR). (Study P05073)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05073
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2010-04-05 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Mometasone Furoate Nasal Spray (MFNS) (Experimental): MFNS 200 mcg total dose (2 sprays each nostril)
  Interventions: Drug: Mometasone Furoate Nasal Spray
- Placebo (Placebo Comparator): Placebo (2 sprays each nostril)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray — Mometasone Furoate Nasal Spray: 2 sprays (50 mcg) each nostril (total 200 mcg)
  Other Names: SCH 032088
  Arms: Mometasone Furoate Nasal Spray (MFNS)
Other: Placebo — Placebo: 2 sprays in each nostril
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well mometasone furoate nasal spray (MFNS) works to relieve SAR symptoms compared to Placebo when symptoms are induced in a chamber setting. Evaluation will be based on subjects self-assessed nose symptoms. Other areas the study will evaluate are: 1) changes in eye symptoms (ocular symptom severity score) after dosing 2) how long MFNS works in relieving the nose (nasal) and eye (ocular) symptoms after 7 daily doses, 3) measurements of nose (nasal) blockage (obstruction), and 4) measurements of the subject's opinion of the study drugs by asking different questions. This study is could last up to 53 days for some subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and to adhere to dose and visit schedules
* 18 to 65 years, either sex, any race
* 2-year history of SAR, being symptomatic during the last 2 ragweed seasons
* Skin test positive to short ragweed allergen at screening, or positive within 12 months
* Women must practice adequate contraception: Females of childbearing potential (including women who are less than 1 year postmenopausal and women who will be sexually active during the study) must agree to use a medically accepted method of contraception or be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Women who are postmenopausal for >1 year (ie, women who have experienced 12 consecutive months of amenorrhea) will be exempted from the use of contraception during the study.; Acceptable methods of contraception include condoms (male and female) with or without a spermicidal agent, diaphragm or cervical cap with a spermicidal agent, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptives, and surgical sterilization (eg, hysterectomy or tubal ligation)
* Negative pregnancy tests during study

Exclusion Criteria:

* Compromised ability to provide informed consent
* Nasal abnormalities, including large nasal polyps, and marked septum deviation that interferes with nasal airflow at screening
* Recent (within the last 2 weeks) or unhealed nasal septum ulcers, nasal surgery, or nasal trauma
* Unstable asthma which cannot be controlled with inhaled short-acting beta-2 agonists
* Diagnosed with sinusitis within the previous 2 weeks
* Is initiating or is currently on advanced immunotherapy
* If on immunotherapy (desensitization therapy), the subject must be stable and should not receive an increase in dose during the study. Subjects may not receive desensitization treatment within 24 hours prior to a study visit
* Is currently on or has been on an antihistamine, decongestant (topical or systemic) or a nasal inhaled corticosteroid during the 14 days prior to the first priming visit
* Unable to refrain from regular use of nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids
* Failed the designated washout periods for any of the prohibited medications
* Upper or lower respiratory tract or sinus infection that required antibiotic therapy or a viral upper or lower respiratory infection within 14 days prior to screening
* Is allergic to or has sensitivity to the study drug or its excipients
* Used any investigational product within 30 days before enrollment or any antibodies for asthma or allergic rhinitis in the past 90 days
* Subject has Chronic obstructive pulmonary disease, Alcohol abuse, Rhinitis medicamentosa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2007-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

REFERENCES:
- [Result] Salapatek AM, Patel P, Gopalan G, Varghese ST. Mometasone furoate nasal spray provides early, continuing relief of nasal congestion and improves nasal patency in allergic patients. Am J Rhinol Allergy. 2010 Nov-Dec;24(6):433-8. doi: 10.2500/ajra.2010.24.3548. Epub 2010 Nov 10. PMID 21067660

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray Day 1: Mometasone Furoate Nasal Spray (MFNS): 2 sprays each nostril (total 200 mcg) for 1 dose
- Placebo Day 1: Placebo: 2 sprays each nostril for 1 dose
- Mometasone Furoate Nasal Spray Day 8: Mometasone Furoate Nasal Spray (MFNS): 2 sprays each nostril (200 mcg daily) for 7 days
- Placebo Day 8: Placebo: 2 sprays each nostril for 7 days
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray Day 1 | Placebo Day 1 | Mometasone Furoate Nasal Spray Day 8 | Placebo Day 8
Started | 77 (All subjects who received MFNS only on Day 1) | 78 (All subjects who received placebo only on Day 1) | 78 (All subjects who received MFNS on Day 1 through Day 7) | 77 (All subjects who received placebo on Day 1 through Day 7)
Completed | 77 | 77 | 74 | 73
Not Completed | 0 | 1 | 4 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray Day 1 | Placebo Day 1 | Mometasone Furoate Nasal Spray Day 8 | Placebo Day 8 | Total
Number analyzed (Participants) | 77 | 78 | 78 | 77 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.1) | 36.3 (10.1) | 36.9 (10.2) | 38.9 (11.2) | 37.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 40 | 44 | 175
  Male | 32 | 32 | 38 | 33 | 135

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Total Nasal Symptom Severity Score (TNSS) at 6 Hours After Dosage Administration on Day 1
Description: Value at 6 hours after dosage administration (Day 1) minus value at Baseline. Minimum threshold TNSS response defined as TNSS score ≥6 out of a possible 12 for combined nasal symptoms of congestion, sneezing, rhinorrhea & itching with a score ≥2 for nasal congestion. Rating of the severity of the individual signs/symptoms according to the following scale: 0=None, sign/symptom wasn't present; 1=Mild, sign/symptom was present, but not disturbing; 2=Moderate, sign/symptom definitely present, & disturbing some of the time; 3=Severe: sign/symptom very noticeable & very bothersome most of the time.
Time Frame: Baseline and 6 hours following initial dosing
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Mometasone Furoate Nasal Spray 200 mcg: All subjects who received 2 sprays each nostril (total 200 mcg) of Mometasone Furoate Nasal Spray (MFNS) on Day 1
- Placebo: All subjects who received 2 sprays each nostril of placebo on Day 1
Arm/Group | Mometasone Furoate Nasal Spray 200 mcg | Placebo
Number analyzed (Participants) | 155 | 155
score on a scale | -2.01 (0.23) | -1.86 (0.23)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray 200 mcg vs Placebo; Test type: Superiority or Other; p = 0.625, ANCOVA; An analysis of covariance (ANCOVA) model was used with treatment as effect and Baseline as a covariate

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray Day 1 | Placebo Day 1 | Mometasone Furoate Nasal Spray Day 8 | Placebo Day 8
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78 | 0/78 | 0/77
Other Adverse Events (participants affected / at risk) | 1/77 | 1/78 | 6/78 | 4/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray Day 1 (N=77) | Placebo Day 1 (N=78) | Mometasone Furoate Nasal Spray Day 8 (N=78) | Placebo Day 8 (N=77)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's represnetatives will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.